CLINICAL TRIAL: NCT04657341
Title: Sonazoid Contrast-enhanced Ultrasound in Assessing Effectiveness of Neoadjuvant Chemotherapy in Breast Cancer Patients.
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Ping Liang, Chief physician, Chinese PLA General Hospital
Other Study IDs: S2020-300-01
Record Dates: First submitted 2020-09-26; First posted 2020-12-08 (Actual); Last update posted 2020-12-08 (Actual); Status verified 2020-12

CONDITIONS: Ultrasound
Keywords: breast

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Sonazoid as a new generation of ultrasound contrast agent.This study based on the features of Sonazoid specific angiography and high mechanical index,the role of Sonazoid in assessing effectiveness of neoadjuvant chemotherapy in breast cancer patients was explored.

DETAILED DESCRIPTION:
This is a prospective, multicenter study.More than 1000 participants will enrolled.Most of them with CEUS,MRI and pathological follow up.When enhanced MRI is needed in the neoadjuvant cycle of patients, Sonazoid-CEUS examination is added at this time point, and postoperative pathology will be used as the gold standard, so as to compare the ability of the two imaging examinations in judging the effect of neoadjuvant chemotherapy.

Investigators will also record the parameter information of imaging examination, pathological type of pathological examination and immunohistochemical index, etc.Contrast-enhanced ultrasound includes lesion location, initial peak tumor volume, 1-minute tumor volume, 2-minute tumor volume, and 5-minute tumor volume, as well as the time for contrast enhancement, contrast agent clearance, and contrast agent clearance.Whether there is no enhancement area in the lesion after contrast enhancement, shape after contrast enhancement, edge after contrast enhancement, order of enhancement, uniformity of enhancement, intensity enhancement, pattern of enhancement, clear boundary after contrast enhancement, aspect ratio after contrast enhancement, etc.The magnetic field strength of the equipment is planned to be recorded in the enhanced MRI information, the name of the MRI contrast agent, the lesion location, the size of the lesion, and the scanning performance are enhanced (lump-like enhancement, non-lump-like enhancement, point-like enhancement), time-signal intensity enhancement curve, DWI signal, ADC value, etc.

ELIGIBILITY:
Inclusion Criteria:

* (1) Refer to the guidelines and specifications for diagnosis and treatment of breast cancer, and it is clearly identified as breast cancer by pathological biopsy.
* (2) Plan to implement NAC therapy;
* (3) All patients and their family members signed informed consent forms, which were approved by the hospital medical Ethics Committee

Exclusion Criteria:

* (1) Those who are known to be allergic to ultrasound contrast agents;
* (2)The subject has a history of allergy to eggs or egg products (i.e. skin rash, dyspnea, swelling of the mouth or throat, hypotension or shock, etc.)
* (3) Intolerance to neoadjuvant chemotherapy;
* (4) Poor compliance with chemotherapy treatment;
* (5) Patients who cannot receive contrast agent MRI examination
* (6) Arteriovenous (left and right) shunt patients in the heart and lungs;
* (7) Mental disorders or mental disorders;
* (8)Patients with serious heart disease or lung disease;
* (9)Pet-pregnant, possibly pregnant or lactating;
* (10)In addition, the researcher or the researcher thinks that the patient is not suitable to participate in this study.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who plan neoadjuvant chemotherapy and conform to contrast-enhanced ultrasound, enhanced mri, and surgical indications.
Sampling Method: Probability Sample
Enrollment: 1012 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Sonazoid contrast-enhanced ultrasound in assessing effectiveness of neoadjuvant chemotherapy in breast cancer patients. | 10 months
  Pathology as a gold standard,to compare the diagnostic performance between contrast-enhanced ultrasound and other contrast-enhanced imaging in neoadjuvant chemotherapy in breast cancer patients.

CONTACTS AND LOCATIONS:
Overall Officials: Ping Liang, Doctor, Principal Investigator — Chinese PLA General Hospital
Locations (1):
- Chinese PLA General Hospital, Beijing, Beijing Municipality, China